CLINICAL TRIAL: NCT00855153
Title: A Pilot Study Using Gradual Virtual Reality Exposure Therapy and D-Cycloserine (DCS) for Treatment of Combat Related Psychological Trauma in Burn Service Members
Brief Title: Virtual Reality and D-Cycloserine in Combat Related Psycological Trauma in Burn Service Members
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator was not able to maintain IRB approval. Study never accrued subjects.
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-09-012
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Psychological Trauma
Keywords: PTSD; burns; virtual reality exposure; D-Cycloserine; Combat related psychological trauma in burned servicemembers
MeSH Terms: conditions — Psychological Trauma; Stress Disorders, Post-Traumatic; Burns | interventions — Cycloserine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): Subjects receive 50mg DCS prior to 90 min session with graded VRE treatment
  Interventions: Other: VR (Virtual reality); Drug: D-Cycloserine

INTERVENTIONS:
Other: VR (Virtual reality) — VR stimulation of combat scenarios utilized as the exposure therapy tool.
  Other Names: Iraq world II
Drug: D-Cycloserine — 50 mg DCS 30 min prior to individual 90 min session with graded VR exposure treatment
  Other Names: DCS

SUMMARY:
The purpose of this pilot study is to begin the examination of the feasibility of using Gradual Virtual Reality Exposure Therapy and D-Cycloserine (DCS) in the management of posttraumatic psychological symptoms in burned OIF/OEF military combatants.

The purpose of a feasibility study is to determine if there is clinical utility in this proposed treatment and to establish effective and safe treatment procedures. Given current literature, the following hypotheses are generated:

Hypothesis 1: Virtual Reality Exposure and D-Cycloserine medication (VRE + DCS learning pill) will result in clinically meaningful PTSD symptom reduction.

1. SMs will attain scores that are lower than initial measures for symptoms of PTSD
2. By the completion of VRE, Ss will attain scores in the sub-clinical range for measures of clinical depression Hypothesis 2: SMs will report greater life satisfaction following completion of VR+DCS treatment, as measured by scores on the Quality of Life Inventory (QOLI) when compared to pre-treatment scores

DETAILED DESCRIPTION:
The purpose of this study is to establish systematic observations about the feasibility of using gradual exposure virtual reality treatment and D-Cycloserine (VRE + DCS) with service members receiving medical care for burns attained during combat. The rational for this study comes from the need to establish with this population, when and how VRE + DCS might be delivered in a safe and systematic fashion. This would be done in preparation for the potential of a future controlled study to address the efficacy of VRE + DCS in comparison to each component and control group.

This study seeks to establish methods of applying VRE + DCS in relation to medical viability as an attempt to clarify at what stage of medical care a service member is able to give informed consent, follow the proscribed instructions, and participate in VRE+ DCS process to include reasonable attention and capacity for immersion. Other areas that will be examined include medication suitability, expected course of medical treatment that would allow for reasonable completion of twelve sessions within twenty weeks, and assessed stability in social support.

ELIGIBILITY:
Inclusion Criteria:

* You are an active duty military male or female service member 18-45 years old and able to participate for duration of care (estimated 12 weeks for initial examination to completion of treatment)
* You have a diagnosis of Post Traumatic Stress Disorder (PTSD) based on a structured clinical interview
* You have a score of greater than 40 on the Clinician Administered PTSD Scale (CAPS)

Exclusion Criteria:

* Psychotic disorders such as schizophrenia, bipolar affective disorder, or history of disruptive non-compliant behaviors
* Borderline intellectual functioning and attention memory problems as identified by standard USAISR neuropsychological screenings;
* Major neurological or major medical difficulties, to include epilepsy/seizures or significant cardiovascular conditions such as heart or blood problems that would be dysregulated by increased anxiety exposure;
* Dependent on drugs based upon screening, self-report or medical record;
* Motion sickness as seen on the VR assessment trial.
* Subjects screened with CAPS scores 44 or lower at pre-treatment assessment.
* Women who are pregnant or breast feeding.
* Unhealed uncovered wounds on face that would be a significant discomfort or infection risk
* Open uncovered wound to hands or face that the doctor sees at being a moderate or greater risk for treatment complications.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Reduction in PTSD symptoms for burn patients and improve perceived life satifaction. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Gaylord, RN, PhD, Principal Investigator — US Army Institute of Surgical Research
Locations (1):
- US Army Institute of Surgical Research, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Davis M, Ressler K, Rothbaum BO, Richardson R. Effects of D-cycloserine on extinction: translation from preclinical to clinical work. Biol Psychiatry. 2006 Aug 15;60(4):369-75. doi: 10.1016/j.biopsych.2006.03.084. PMID 16919524